CLINICAL TRIAL: NCT07372001
Title: Effects on Facial Skin Aging After Topical Application of Exosomes With a Microneedling Device
Acronym: EFSATAEMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2024/04/02
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Skin Aging
Keywords: Exosomes.; Skin; Skin Aging; Rejuvenation

STUDY DESIGN:
Intervention Model Description: This was a clinical, experimental, prospective, and comparative investigation conducted in a before-and-after format
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical lyophilized exosomes application (Other): The exosomes were applied to the facial area by dripping onto the skin and using a microneedling device to enhance dermal penetration. Three sessions, each four weeks apart, were performed for each subject.
  Interventions: Biological: Topical lyophilized exosomes application

INTERVENTIONS:
Biological: Topical lyophilized exosomes application — The exosomes were applied to the facial area by dripping onto the skin and using a microneedling device to enhance dermal penetration. Three sessions, each four weeks apart, were performed for each subject
  Other Names: Exosomes

SUMMARY:
In this study, we evaluated the extent of reversal of facial dermal aging signs using topical lyophilized exosomes with a microneedling device

DETAILED DESCRIPTION:
This clinical, experimental, prospective, and comparative investigation was conducted in a before-and-after format. The exosomes were applied to the facial area by dripping onto the skin and using a microneedling device to enhance dermal penetration. Three sessions, each four weeks apart, were performed for each subject. During each session, documentation was performed using photographs and the SAASQ and FaceQ visual scales for objective and subjective evaluations, respectively. ANOVA test for repeated measures was used for the statistical analysis. SPSS version 31.0 was used for the analysis.

All measured variables, both objective and subjective, were favorable for the use of exosomes as a treatment for early signs of aging.

This pilot study provides preliminary results showing an excellent cosmetic response to exosome treatment using microneedling, with good user satisfaction and tolerable and harmless adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 50 with facial rhytides and a minimum score of 12 on the SASSQ scale

Exclusion Criteria:

* pregnancy or breastfeeding, active acne or rosacea, local infections, lesions suspicious for malignancy, and allergy to exosomes. The elimination criteria involved loss of follow-up of the research subject and the occurrence of an allergic reaction or intolerable adverse effects.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Facial dermal changes | From enrollment to the end of treatment at 8 weeks
  Six skin characteristics were evaluated using SASSQ visual scale: elasticity, wrinkles, roughness, pigmentation, erythema, and pore size
Subjective evaluation of facial dermal changes | From enrollment to the end of treatment at 8 weeks
  The FACE-Q Aesthetics questionnaire was utilized, comprising 37 independent functional scales and six checklists that measure patient-relevant outcomes from their perspective. In this study, the following scales from this questionnaire were used: expectations (before), satisfaction with skin (before and after), psychosocial distress related to appearance (before and after), assessment of facial lines: general impression (before and after), and satisfaction with the decision (after). Additionally, an adverse effects scale was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología F.A.P. Conde de Valenciana, I.A.P., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: March 2026 - June 2026

REFERENCES:
- [Result] Kieser M, Wassmer G. On the use of the upper confidence limit for the variance from a pilot sample for sample size determination. Biom J. 1996;38(8):941-9. doi: 10.1002/bimj.4710380806
- [Result] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Result] Alzahrani FA. Melatonin improves therapeutic potential of mesenchymal stem cells-derived exosomes against renal ischemia-reperfusion injury in rats. Am J Transl Res. 2019 May 15;11(5):2887-2907. eCollection 2019. PMID 31217862
- [Result] Shin KO, Ha DH, Kim JO, Crumrine DA, Meyer JM, Wakefield JS, Lee Y, Kim B, Kim S, Kim HK, Lee J, Kwon HH, Park GH, Lee JH, Lim J, Park S, Elias PM, Park K, Yi YW, Cho BS. Exosomes from Human Adipose Tissue-Derived Mesenchymal Stem Cells Promote Epidermal Barrier Repair by Inducing de Novo Synthesis of Ceramides in Atopic Dermatitis. Cells. 2020 Mar 10;9(3):680. doi: 10.3390/cells9030680. PMID 32164386
- [Result] Hu S, Li Z, Cores J, Huang K, Su T, Dinh PU, Cheng K. Needle-Free Injection of Exosomes Derived from Human Dermal Fibroblast Spheroids Ameliorates Skin Photoaging. ACS Nano. 2019 Oct 22;13(10):11273-11282. doi: 10.1021/acsnano.9b04384. Epub 2019 Aug 26. PMID 31449388
- [Result] Liu M, Wang H, Liu Z, Liu G, Wang W, Li X. Exosomes from adipose-derived stem cells inhibits skin cancer progression via miR-199a-5p/SOX4. Biotechnol Genet Eng Rev. 2024 Dec;40(4):3950-3962. doi: 10.1080/02648725.2023.2204702. Epub 2023 Apr 24. PMID 37092869
- [Result] Lueangarun S, Cho BS, Tempark T. Topical moisturizer with rose stem cell-derived exosomes (RSCEs) for recalcitrant seborrheic dermatitis: A case report with 6 months of follow-up. J Cosmet Dermatol. 2024 Oct;23(10):3128-3132. doi: 10.1111/jocd.16389. Epub 2024 Jun 3. PMID 38831604
- [Result] Hade MD, Suire CN, Suo Z. Mesenchymal Stem Cell-Derived Exosomes: Applications in Regenerative Medicine. Cells. 2021 Aug 1;10(8):1959. doi: 10.3390/cells10081959. PMID 34440728
- [Result] Ha DH, Kim HK, Lee J, Kwon HH, Park GH, Yang SH, Jung JY, Choi H, Lee JH, Sung S, Yi YW, Cho BS. Mesenchymal Stem/Stromal Cell-Derived Exosomes for Immunomodulatory Therapeutics and Skin Regeneration. Cells. 2020 May 7;9(5):1157. doi: 10.3390/cells9051157. PMID 32392899
- [Result] 6. Ma J, Yong L, Lei P, Li H, Fang Y, Wang L, et al. Advances in microRNA from adipose-derived mesenchymal stem cell-derived exosome: focusing on wound healing. J Mater Chem B Mater Biol Med. 2022;10(46):9565-77. doi: 10.1039/D2TB01987F
- [Result] Ottenhof MJ, Veldhuizen IJ, Hensbergen LJV, Blankensteijn LL, Bramer W, Lei BV, Hoogbergen MM, Hulst RRWJ, Sidey-Gibbons CJ. The Use of the FACE-Q Aesthetic: A Narrative Review. Aesthetic Plast Surg. 2022 Dec;46(6):2769-2780. doi: 10.1007/s00266-022-02974-9. Epub 2022 Jun 28. PMID 35764813
- [Result] Eiben-Nielson C, Kerscher M. Development and validation of a global photonumeric scale for evaluating skin quality of aged female facial skin. J Cosmet Dermatol. 2021 Dec;20(12):4032-4039. doi: 10.1111/jocd.14058. Epub 2021 Mar 24. PMID 33690945
- [Result] Rorteau J, Chevalier FP, Fromy B, Lamartine J. [Functional integrity of aging skin, from cutaneous biology to anti-aging strategies]. Med Sci (Paris). 2020 Dec;36(12):1155-1162. doi: 10.1051/medsci/2020223. Epub 2020 Dec 9. French. PMID 33296632
- [Result] Csekes E, Rackova L. Skin Aging, Cellular Senescence and Natural Polyphenols. Int J Mol Sci. 2021 Nov 23;22(23):12641. doi: 10.3390/ijms222312641. PMID 34884444
- [Result] Kanitakis J. Anatomy, histology and immunohistochemistry of normal human skin. Eur J Dermatol. 2002 Jul-Aug;12(4):390-9; quiz 400-1. PMID 12095893